CLINICAL TRIAL: NCT00475852
Title: Double-Blind, Placebo-Controlled, Multicenter Acute Study of Clinical Effectiveness of Nesiritide in Subjects With Decompensated Heart Failure (ASCEND-HF)
Brief Title: A Study Testing the Effectiveness of Nesiritide in Patients With Acute Decompensated Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR013954; ASCEND-HF (Other: Johnson & Johnson Pharmaceutical Research & Development, LLC); A093 (Other: Johnson & Johnson Pharmaceutical Research & Development, LLC); NATRECORAHF3002 (Other: Johnson & Johnson Pharmaceutical Research & Development, LLC)
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Results first posted 2012-05-10 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Heart Decompensation
Keywords: Heart Decompensation; Dyspnea; Heart failure; Nesiritide; Decompensated; ADHF
MeSH Terms: conditions — Heart Failure; Dyspnea | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Nesiritide 0.01 mcg/kg/min intravenous (IV) infusion (with or without 2 mcg/kg bolus) for 24 to 168 hours (hrs)
  Interventions: Drug: Nesiritide
- 002 (Placebo Comparator): Placebo matching placebo infusion:0.01 mcg/kg/min IV infusion (with or without 2 mcg/kg bolus) for 24 to 168 hrs
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nesiritide — 0.01 mcg/kg/min IV infusion (with or without 2 mcg/kg bolus) for 24 to 168 hrs
  Arms: 001
Drug: Placebo — matching placebo infusion:0.01 mcg/kg/min IV infusion (with or without 2 mcg/kg bolus) for 24 to 168 hrs
  Arms: 002

SUMMARY:
The purpose of this study is to find out if nesiritide (a human B-type natriuretic peptide/hBNP) as compared to placebo, plus the usual treatment for acute decompensated heart failure, helps to improve breathing difficulties, reduce heart failure readmissions to hospitals, and helps patients live longer.

DETAILED DESCRIPTION:
Acute Decompensated Heart Failure (ADHF) is the inability of the heart to pump efficiently, which can result in symptoms like shortness of breath at rest or with minimal activity. ADHF is a condition in which the heart cannot perform the necessary circulation of blood through the body. This is a randomized (study medication is assigned by chance), double-blind (neither the patient or the doctor knows whether the patient is assigned to receive study drug or placebo [does not contain study drug]), placebo-controlled, parallel group, multicenter study of the effectiveness of nesiritide administered continuously through a vein for a minimum of 24 hours up to a maximum of 7 days. The study hypothesis is that nesiritide given in addition to standard care is superior to placebo given in addition to standard care as measured by relief of breathing difficulties (by patient evaluation utilizing a breathlessness scale) at 6 hours or 24 hours after nesiritide administration, and reduction in rehospitalization due to heart failure and death from study drug administration through Day 30. The study drug (nesiritide) or placebo dose being studied is 0.010 mcg/kg/min with or without a 2 mcg/kg initial bolus (one time injection) of nesiritide. Patient safety will be monitored throughout the study through physical exams, vital signs (heart rate, blood pressure, respiratory rate, and temperature), blood tests, and side effects. The patients assigned to the nesiritide group will receive a continuous intravenous (into a vein) infusion at 0.010 mcg/kg/min of nesiritide with or without a 2 mcg/kg bolus (one time injection). The patients assigned to the placebo group will receive matching placebo bolus and infusion. The bolus is given over one minute and the continuous infusion is given for at least 24 hours and up to 7 days.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized for the management of acute decompensated heart failure (ADHF) or diagnosed with ADHF within 48 hours after being hospitalized for another reason; Diagnosis of ADHF is defined as dyspnea (difficulty breathing) at rest or dyspnea with minimal activity.

Exclusion Criteria:

At high risk for hypotension (low blood pressure); Acute coronary syndrome as primary diagnosis; History of cardiac valvular stenosis, restrictive cardiomyopathy, hypertrophic cardiomyopathy, or pericardial tamponade; Previous enrollment in a nesiritide study; Persistent, uncontrolled hypertension (SBP [systolic blood pressure] >180 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7141 (Actual)
Dates: Start 2007-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.
Locations (328):
- United States (171):
  - Huntsville, Alabama
  - Mobile, Alabama
  - Anchorage, Alaska
  - Gilbert, Arizona
  - Scottsdale, Arizona
  - Fort Smith, Arkansas
  - Jonesboro, Arkansas
  - Berkeley, California
  - Culver City, California
  - Escondido, California
  - Inglewood, California
  - Loma Linda, California
  - Los Angeles, California
  - Mission Viejo, California
  - Sacramento, California
  - San Diego, California
  - Santa Ana, California
  - Torrance, California
  - Ventura, California
  - Denver, Colorado
  - Englewood, Colorado
  - Fort Collins, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Fort Lauderdale, Florida
  - Gainesville, Florida
  - Inverness, Florida
  - Lakeland, Florida
  - Melbourne, Florida
  - Miami Beach, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Gainesville, Georgia
  - Macon, Georgia
  - Aurora, Illinois
  - Chicago, Illinois
  - Downers Grove, Illinois
  - Elk Grove Village, Illinois
  - Hinsdale, Illinois
  - La Grange, Illinois
  - Maywood, Illinois
  - Mokena, Illinois
  - Oakbrook Terrace, Illinois
  - Peoria, Illinois
  - Rockford, Illinois
  - Springfield, Illinois
  - Anderson, Indiana
  - Indianapolis, Indiana
  - Munster, Indiana
  - South Bend, Indiana
  - Valparaiso, Indiana
  - Danville, Kentucky
  - Edgewood, Kentucky
  - Lexington, Kentucky
  - Owensboro, Kentucky
  - Baltimore, Maryland
  - Randallstown, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Brighton, Massachusetts
  - Springfield, Massachusetts
  - Worcester, Massachusetts
  - Bay City, Michigan
  - Detroit, Michigan
  - Flint, Michigan
  - Lansing, Michigan
  - Monroe, Michigan
  - Petoskey, Michigan
  - Pontiac, Michigan
  - Saginaw, Michigan
  - Troy, Michigan
  - Minneapolis, Minnesota
  - Tupelo, Mississippi
  - Kansas City, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Papillion, Nebraska
  - Manchester, New Hampshire
  - Browns Mills, New Jersey
  - Camden, New Jersey
  - Elmer, New Jersey
  - Hackensack, New Jersey
  - Neptune City, New Jersey
  - Newark, New Jersey
  - Paterson, New Jersey
  - Ridgewood, New Jersey
  - Toms River, New Jersey
  - Trenton, New Jersey
  - Turnersville, New Jersey
  - Albany, New York
  - Brooklyn, New York
  - Elmhurst, New York
  - Johnson City, New York
  - New Hyde Parke, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Roslyn, New York
  - Saratoga Springs, New York
  - Stony Brook, New York
  - The Bronx, New York
  - Valhalla, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Gastonia, North Carolina
  - Greenville, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Garfield Heights, Ohio
  - Mansfield, Ohio
  - Mayfield Heights, Ohio
  - Middletown, Ohio
  - Sylvania, Ohio
  - Toledo, Ohio
  - Youngstown, Ohio
  - Midwest City, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Bend, Oregon
  - Abington, Pennsylvania
  - Allentown, Pennsylvania
  - Beaver, Pennsylvania
  - Bethlehem, Pennsylvania
  - Camp Hill, Pennsylvania
  - Danville, Pennsylvania
  - Harrisburg, Pennsylvania
  - Lancaster, Pennsylvania
  - Natrona Heights, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - York, Pennsylvania
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Spartanburg, South Carolina
  - Sumter, South Carolina
  - Rapid City, South Dakota
  - Kingsport, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Oak Ridge, Tennessee
  - Amarillo, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Tyler, Texas
  - Falls Church, Virginia
  - Harrisonburg, Virginia
  - Lynchburg, Virginia
  - Norfolk, Virginia
  - Winchester, Virginia
  - Tacoma, Washington
  - Burlington, Wisconsin
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Argentina (6):
  - Buenos Aires
  - Córdoba
  - La Plata
  - Mar del Plata
  - San Miguel de Tucumán
  - Santa Fe
- Australia (11):
  - Bedford
  - Camperdown
  - Concord
  - Darlinghurst
  - Elizabeth Vale
  - Fitzroy
  - Hobart
  - Kogarah
  - Launceston
  - Melbourne
  - Randwick
- Brazil (11):
  - Belo Horizonte
  - Campinas
  - Curitiba
  - Fortaleza
  - Goiânia
  - Porto Alegre
  - Recife
  - Rio de Janeiro-Rj
  - Salvador
  - São José do Rio Preto
  - São Paulo
- Bulgaria (3):
  - Pleven
  - Sofia
  - Varna
- Canada (28):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Red Deer, Alberta
  - Campbell River, British Columbia
  - Kelowna, British Columbia
  - Maple Ridge, British Columbia
  - New Westminster, British Columbia
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Lakeland, Manitoba
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Ajax, Ontario
  - Brampton, Ontario
  - Cornwall, Ontario
  - Hamilton, Ontario
  - Kitchener, Ontario
  - Ottawa, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Granby, Quebec
  - Laval, Quebec
  - Montreal, Quebec
  - Saint-Charles-Borromée, Quebec
  - Sherbrooke, Quebec
  - Ste-Foy, Quebec
  - Terrebonne, Quebec
- Chile (3):
  - Santiago
  - Santiago Rm
  - Temuco
- China (8):
  - Beijing
  - Beijing Prc
  - Guangdong Province
  - Hangzhou
  - Jinan
  - Shanghai
  - Tianjin
  - Xi'an
- Colombia (3):
  - Barranquilla
  - Bogotá Dc
  - Floridablanca
- France (8):
  - Colmar
  - Paris
  - Poitiers
  - Pontoise
  - Thionville Cedex N/A
  - Toulouse
  - Valenciennes
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Bad Krozingen
  - Berlin
  - Brandenburg
  - Ludwigshafen
  - Lüdenscheid
  - Neuruppin
- Greece (4):
  - Athens
  - Larissa
  - Thessalonikis
  - Volos
- India (7):
  - Ahmedabad
  - Bengaluru
  - Coimbatore
  - Hyderabad
  - Nagpur
  - Pune
  - Vadodara
- Israel (6):
  - Hadera
  - Haifa
  - Holon
  - Petah Tikva
  - Ramat Gan
  - Safed
- Lithuania (2):
  - Kaunas
  - Vilnius Lt
- Malaysia (2):
  - Johor Bahru
  - Kuala Lumpur
- Mexico (5):
  - Aguascalientes
  - Guadalajara
  - San Luis Potosí City
  - Sinaloa
  - Zapopan
- Netherlands (6):
  - Amersfoort
  - Delft
  - Gorinchem
  - Groningen
  - Leeuwarden
  - Sneek
- New Zealand (6):
  - Auckland
  - Christchurch
  - Hamilton
  - Hastings
  - Lower Hutt
  - Nelson
- Norway (3):
  - Stavanger
  - Trondheim
  - Tønsberg
- Poland (7):
  - Bydgoszcz
  - Gdynia
  - Krakow
  - Ostrowiec Świętokrzyski
  - Skierniewice
  - Warsaw
  - Wroclaw
- Russia (5):
  - Kemerovo
  - Moscow
  - Tomsk
  - Tyumen
  - Yekaterinburg
- Singapore, Singapore
- South Korea (2):
  - Chungcheongbuk-Do
  - Seoul
- Sweden (2):
  - Falun
  - Uppsala
- Taiwan (3):
  - Kaohsiung City
  - Taipei
  - Taoyuan District
- Thailand (2):
  - Bangkok
  - Khon Kaen
- Ukraine (7):
  - Dnipro
  - Donetsk
  - Kharkiv
  - Lviv
  - Mykolayiv
  - Vinnitsa
  - Zaporizhzhya

REFERENCES:
- [Derived] Gui H, Tang WHW, Francke S, Li J, She R, Bazeley P, Pereira NL, Adams K, Luzum JA, Connolly TM, Hernandez AF, McNaughton CD, Williams LK, Lanfear DE. Common Variants on FGD5 Increase Hazard of Mortality or Rehospitalization in Patients With Heart Failure From the ASCEND-HF Trial. Circ Heart Fail. 2023 Sep;16(9):e010438. doi: 10.1161/CIRCHEARTFAILURE.122.010438. Epub 2023 Jul 26. PMID 37725680
- [Derived] Cosiano MF, Vista A, Sun JL, Alhanti B, Harrington J, Butler J, Starling RC, Mentz RJ, Greene SJ. Comparing New York Heart Association Class and Patient-Reported Outcomes Among Patients Hospitalized for Heart Failure. Circ Heart Fail. 2023 Jan;16(1):e010107. doi: 10.1161/CIRCHEARTFAILURE.122.010107. Epub 2022 Oct 31. PMID 36314126
- [Derived] Blumer V, Mentz RJ, Sun JL, Butler J, Metra M, Voors AA, Hernandez AF, O'Connor CM, Greene SJ. Prognostic Role of Prior Heart Failure Hospitalization Among Patients Hospitalized for Worsening Chronic Heart Failure. Circ Heart Fail. 2021 Apr;14(4):e007871. doi: 10.1161/CIRCHEARTFAILURE.120.007871. Epub 2021 Mar 29. PMID 33775110
- [Derived] Greene SJ, DeVore AD, Sheng S, Fonarow GC, Butler J, Califf RM, Hernandez AF, Matsouaka RA, Samman Tahhan A, Thomas KL, Vaduganathan M, Yancy CW, Peterson ED, O'Connor CM, Mentz RJ. Representativeness of a Heart Failure Trial by Race and Sex: Results From ASCEND-HF and GWTG-HF. JACC Heart Fail. 2019 Nov;7(11):980-992. doi: 10.1016/j.jchf.2019.07.011. Epub 2019 Oct 9. PMID 31606362
- [Derived] Greene SJ, Hernandez AF, Sun JL, Butler J, Armstrong PW, Ezekowitz JA, Zannad F, Ferreira JP, Coles A, Metra M, Voors AA, Califf RM, O'Connor CM, Mentz RJ. Relationship Between Enrolling Country Income Level and Patient Profile, Protocol Completion, and Trial End Points. Circ Cardiovasc Qual Outcomes. 2018 Oct;11(10):e004783. doi: 10.1161/CIRCOUTCOMES.118.004783. PMID 30354576
- [Derived] Verma AK, Sun JL, Hernandez A, Teerlink JR, Schulte PJ, Ezekowitz J, Voors A, Starling R, Armstrong P, O'Conner CM, Mentz RJ. Rate pressure product and the components of heart rate and systolic blood pressure in hospitalized heart failure patients with preserved ejection fraction: Insights from ASCEND-HF. Clin Cardiol. 2018 Jul;41(7):945-952. doi: 10.1002/clc.22981. Epub 2018 Jul 17. PMID 29781109
- [Derived] Bhatt AS, Cooper LB, Ambrosy AP, Clare RM, Coles A, Joyce E, Krishnamoorthy A, Butler J, Felker GM, Ezekowitz JA, Armstrong PW, Hernandez AF, O'Connor CM, Mentz RJ. Interaction of Body Mass Index on the Association Between N-Terminal-Pro-b-Type Natriuretic Peptide and Morbidity and Mortality in Patients With Acute Heart Failure: Findings From ASCEND-HF (Acute Study of Clinical Effectiveness of Nesiritide in Decompensated Heart Failure). J Am Heart Assoc. 2018 Feb 3;7(3):e006740. doi: 10.1161/JAHA.117.006740. PMID 29431103
- [Derived] Greene SJ, Hernandez AF, Dunning A, Ambrosy AP, Armstrong PW, Butler J, Cerbin LP, Coles A, Ezekowitz JA, Metra M, Starling RC, Teerlink JR, Voors AA, O'Connor CM, Mentz RJ. Hospitalization for Recently Diagnosed Versus Worsening Chronic Heart Failure: From the ASCEND-HF Trial. J Am Coll Cardiol. 2017 Jun 27;69(25):3029-3039. doi: 10.1016/j.jacc.2017.04.043. PMID 28641792
- [Derived] Greene SJ, Hernandez AF, Sun JL, Metra M, Butler J, Ambrosy AP, Ezekowitz JA, Starling RC, Teerlink JR, Schulte PJ, Voors AA, Armstrong PW, O'Connor CM, Mentz RJ. Influence of Clinical Trial Site Enrollment on Patient Characteristics, Protocol Completion, and End Points: Insights From the ASCEND-HF Trial (Acute Study of Clinical Effectiveness of Nesiritide in Decompensated Heart Failure). Circ Heart Fail. 2016 Sep;9(9):e002986. doi: 10.1161/CIRCHEARTFAILURE.116.002986. PMID 27623769
- [Derived] Ezekowitz JA, Podder M, Hernandez AF, Armstrong PW, Starling RC, O'Connor CM, Califf RM. Arrival by ambulance in acute heart failure: insights into the mode of presentation from Acute Studies of Nesiritide in Decompensated Heart Failure (ASCEND-HF). BMJ Open. 2016 Mar 17;6(3):e010201. doi: 10.1136/bmjopen-2015-010201. PMID 26988350
- [Derived] Abualnaja S, Podder M, Hernandez AF, McMurray JJ, Starling RC, O'Connor CM, Califf RM, Armstrong PW, Ezekowitz JA. Acute Heart Failure and Atrial Fibrillation: Insights From the Acute Study of Clinical Effectiveness of Nesiritide in Decompensated Heart Failure (ASCEND-HF) Trial. J Am Heart Assoc. 2015 Aug 24;4(8):e002092. doi: 10.1161/JAHA.115.002092. PMID 26304935
- [Derived] Patel PA, Heizer G, O'Connor CM, Schulte PJ, Dickstein K, Ezekowitz JA, Armstrong PW, Hasselblad V, Mills RM, McMurray JJ, Starling RC, Tang WH, Califf RM, Hernandez AF. Hypotension during hospitalization for acute heart failure is independently associated with 30-day mortality: findings from ASCEND-HF. Circ Heart Fail. 2014 Nov;7(6):918-25. doi: 10.1161/CIRCHEARTFAILURE.113.000872. Epub 2014 Oct 3. PMID 25281655
- [Derived] van Deursen VM, Hernandez AF, Stebbins A, Hasselblad V, Ezekowitz JA, Califf RM, Gottlieb SS, O'Connor CM, Starling RC, Tang WH, McMurray JJ, Dickstein K, Voors AA. Nesiritide, renal function, and associated outcomes during hospitalization for acute decompensated heart failure: results from the Acute Study of Clinical Effectiveness of Nesiritide and Decompensated Heart Failure (ASCEND-HF). Circulation. 2014 Sep 16;130(12):958-65. doi: 10.1161/CIRCULATIONAHA.113.003046. Epub 2014 Jul 29. PMID 25074507
- [Derived] Kaul P, Reed SD, Hernandez AF, Howlett JG, Ezekowitz JA, Li Y, Zheng Y, Rouleau JL, Starling RC, O'Connor CM, Califf RM, Armstrong PW. Differences in treatment, outcomes, and quality of life among patients with heart failure in Canada and the United States. JACC Heart Fail. 2013 Dec;1(6):523-30. doi: 10.1016/j.jchf.2013.07.004. Epub 2013 Oct 23. PMID 24622005
- [Derived] Toma M, Ezekowitz JA, Bakal JA, O'Connor CM, Hernandez AF, Sardar MR, Zolty R, Massie BM, Swedberg K, Armstrong PW, Starling RC. The relationship between left ventricular ejection fraction and mortality in patients with acute heart failure: insights from the ASCEND-HF Trial. Eur J Heart Fail. 2014 Mar;16(3):334-41. doi: 10.1002/ejhf.19. Epub 2013 Dec 14. PMID 24464687
- [Derived] Reed SD, Kaul P, Li Y, Eapen ZJ, Davidson-Ray L, Schulman KA, Massie BM, Armstrong PW, Starling RC, O'Connor CM, Hernandez AF, Califf RM. Medical resource use, costs, and quality of life in patients with acute decompensated heart failure: findings from ASCEND-HF. J Card Fail. 2013 Sep;19(9):611-20. doi: 10.1016/j.cardfail.2013.07.003. PMID 24054337
- [Derived] Howlett JG, Ezekowitz JA, Podder M, Hernandez AF, Diaz R, Dickstein K, Dunlap ME, Corbalan R, Armstrong PW, Starling RC, O'Connor CM, Califf RM, Fonarow GC; ASCEND-HF Investigators. Global variation in quality of care among patients hospitalized with acute heart failure in an international trial: findings from the acute study clinical effectiveness of nesiritide in decompensated heart failure trial (ASCEND-HF). Circ Cardiovasc Qual Outcomes. 2013 Sep 1;6(5):534-42. doi: 10.1161/CIRCOUTCOMES.113.000119. Epub 2013 Jul 30. PMID 23899930
- [Derived] Eapen ZJ, Reed SD, Li Y, Kociol RD, Armstrong PW, Starling RC, McMurray JJ, Massie BM, Swedberg K, Ezekowitz JA, Fonarow GC, Teerlink JR, Metra M, Whellan DJ, O'Connor CM, Califf RM, Hernandez AF. Do countries or hospitals with longer hospital stays for acute heart failure have lower readmission rates?: Findings from ASCEND-HF. Circ Heart Fail. 2013 Jul;6(4):727-32. doi: 10.1161/CIRCHEARTFAILURE.112.000265. Epub 2013 Jun 14. PMID 23770519
- [Derived] Ezekowitz JA, Hu J, Delgado D, Hernandez AF, Kaul P, Leader R, Proulx G, Virani S, White M, Zieroth S, O'Connor C, Westerhout CM, Armstrong PW. Acute heart failure: perspectives from a randomized trial and a simultaneous registry. Circ Heart Fail. 2012 Nov;5(6):735-41. doi: 10.1161/CIRCHEARTFAILURE.112.968974. Epub 2012 Oct 2. PMID 23032196
- [Derived] Ezekowitz JA, Hernandez AF, O'Connor CM, Starling RC, Proulx G, Weiss MH, Bakal JA, Califf RM, McMurray JJ, Armstrong PW. Assessment of dyspnea in acute decompensated heart failure: insights from ASCEND-HF (Acute Study of Clinical Effectiveness of Nesiritide in Decompensated Heart Failure) on the contributions of peak expiratory flow. J Am Coll Cardiol. 2012 Apr 17;59(16):1441-8. doi: 10.1016/j.jacc.2011.11.061. PMID 22497823
- [Derived] O'Connor CM, Starling RC, Hernandez AF, Armstrong PW, Dickstein K, Hasselblad V, Heizer GM, Komajda M, Massie BM, McMurray JJ, Nieminen MS, Reist CJ, Rouleau JL, Swedberg K, Adams KF Jr, Anker SD, Atar D, Battler A, Botero R, Bohidar NR, Butler J, Clausell N, Corbalan R, Costanzo MR, Dahlstrom U, Deckelbaum LI, Diaz R, Dunlap ME, Ezekowitz JA, Feldman D, Felker GM, Fonarow GC, Gennevois D, Gottlieb SS, Hill JA, Hollander JE, Howlett JG, Hudson MP, Kociol RD, Krum H, Laucevicius A, Levy WC, Mendez GF, Metra M, Mittal S, Oh BH, Pereira NL, Ponikowski P, Tang WH, Tanomsup S, Teerlink JR, Triposkiadis F, Troughton RW, Voors AA, Whellan DJ, Zannad F, Califf RM. Effect of nesiritide in patients with acute decompensated heart failure. N Engl J Med. 2011 Jul 7;365(1):32-43. doi: 10.1056/NEJMoa1100171. PMID 21732835
- See also: A study testing the effectiveness of Nesiritide in Patients with Acute Decompensated Heart Failure — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=970&filename=CR013954_REF.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Double-Blind, Placebo-Controlled, Multicenter Acute Study of Clinical Effectiveness of Nesiritide in Subjects With Decompensated Heart Failure (ASCEND-HF)
Period: Overall Study
Arm/Group | Nesiritide | Placebo
Started | 3564 | 3577
Completed | 3047 | 3029
Not Completed | 517 | 548
Not completed — Death | 444 | 456
Not completed — Withdrawal by Subject | 19 | 24
Not completed — Lost to Follow-up | 54 | 68

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nesiritide | Placebo | Total
Number analyzed (Participants) | 3564 | 3577 | 7141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 2 | 6
  Between 18 and 65 years | 1572 | 1597 | 3169
  >=65 years | 1988 | 1978 | 3966
Age Continuous [Mean (Standard Deviation); unit: years] | 65.5 (14.09) | 65.4 (14.20) | 65.5 (14.14)
Age, Customized [Number; unit: participants]
  <=64 | 1576 | 1599 | 3175
  65-74 | 938 | 901 | 1839
  >=75 | 1050 | 1077 | 2127
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1197 | 1247 | 2444
  Male | 2367 | 2330 | 4697
Region of Enrollment [Number; unit: participants]
  ARG | 108 | 108 | 216
  AUS | 18 | 16 | 34
  BGR | 35 | 32 | 67
  BRA | 73 | 77 | 150
  CAN | 240 | 236 | 476
  CHL | 25 | 25 | 50
  CHN | 154 | 160 | 314
  COL | 15 | 15 | 30
  DEU | 3 | 3 | 6
  FRA | 51 | 47 | 98
  GRC | 24 | 24 | 48
  IND | 499 | 502 | 1001
  ISR | 38 | 40 | 78
  ITA | 36 | 36 | 72
  KOR | 74 | 74 | 148
  LTU | 48 | 49 | 97
  MEX | 108 | 111 | 219
  MYS | 38 | 37 | 75
  NLD | 71 | 70 | 141
  NOR | 27 | 29 | 56
  NZL | 7 | 7 | 14
  POL | 134 | 133 | 267
  ROU | 24 | 28 | 52
  RUS | 148 | 147 | 295
  SGP | 27 | 26 | 53
  SWE | 2 | 3 | 5
  THA | 23 | 23 | 46
  TWN | 38 | 39 | 77
  UKR | 97 | 92 | 189
  USA | 1379 | 1388 | 2767
Baseline BMI [Mean (Standard Deviation); unit: kg/cm2] | 28.9 (7.86) | 29.1 (7.77) | 29.0 (7.81)

OUTCOME MEASURES:

1. Primary Outcome: Composite of Rehospitalization Due to Heart Failure and All-Cause Mortality
Time Frame: Randomization to Day 30
Population: The modified intent-to-treat (MITT) population consisted of all randomized patients who received any amount of study medication and was the primary analysis population for all efficacy endpoints. 141 and 164 patients in the nesiritide and placebo groups, respectively, were not MITT population eligible or didn't have outcome measure of interest.
Measure: Number; unit: Participants
Groups:
- Placebo: Matching placebo infusion 0.01 mcg/kg/min IV infusion (with or without 2 mcg/kg bolus) for 24 to 168 hrs
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3423 | 3413
Participants | 321 | 345
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p = 0.313, Cochran-Mantel-Haenszel; Stratified by geographical region; Risk Difference (RD) = -0.7, 95% CI 2-sided [-2.1 to 0.7]

2. Primary Outcome: Dyspnea Self-Assessment at 6 Hours After Initiation of Study Drug
Description: Dyspnea symptoms were measured by patient self-assessed Likert scale at 6 hours after study drug initiation.The Likert scale is a 7-point ordinal categorical scale (the 7 categories are markedly better, moderately better, minimally better, unchanged, minimally worse, moderately worse, and markedly worse.)
Time Frame: 6 hours after initiation of study drug
Population: The modified intent-to-treat (MITT) population consisted of all randomized patients who received any amount of study medication and was the primary analysis population for all efficacy endpoints. 148 and 133 patients in the nesiritide and placebo groups, respectively, were not MITT population eligible or didn't have outcome measure of interest.
Measure: Number; unit: Participants
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3416 | 3444
Participants
  Markedly Better | 513 | 460
  Moderately Better | 1007 | 989
  Minimally Better | 1119 | 1174
  No Change | 692 | 748
  Minimally Worse | 39 | 40
  Moderately Worse | 12 | 13
  Markedly Worse | 34 | 20
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p = 0.030, Van Elteren test; Controlled for region

3. Primary Outcome: Dyspnea Self-Assessment at 24 Hours After Initiation of Study Drug
Description: Dyspnea symptoms were measured by patient self-assessed Likert scale at 24 hours after study drug initiation. The Likert scale is a 7-point ordinal categorical scale (the 7 categories are markedly better, moderately better, minimally better, unchanged, minimally worse, moderately worse, and markedly worse.)
Time Frame: 24 hours after study drug initiation
Population: The modified intent-to-treat (MITT) population consisted of all randomized patients who received any amount of study medication and was the primary analysis population for all efficacy endpoints. 193 and 179 patients in the nesiritide and placebo groups, respectively, were not MITT population eligible or didn't have outcome measure of interest.
Measure: Number; unit: Participants
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3371 | 3398
Participants
  Markedly Better | 1025 | 935
  Moderately Better | 1274 | 1313
  Minimally Better | 716 | 751
  No Change | 291 | 323
  Minimally Worse | 27 | 36
  Moderately Worse | 7 | 15
  Markedly Worse | 31 | 25
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p = 0.007, Van Elteren test; Controlled for region

4. Secondary Outcome: Overall Well-Being Self-Assessment at 6 Hours After Initiation of Study Drug
Description: Overall well-being was measured by patient self-assessed Likert scale at 6 hours after study drug initiation. The Likert scale is a 7-point ordinal categorical scale (the 7 categories are markedly better, moderately better, minimally better, unchanged, minimally worse, moderately worse, and markedly worse.)
Time Frame: 6 hours after study drug initiation
Population: The modified intent-to-treat (MITT) population consisted of all randomized patients who received any amount of study medication and was the primary analysis population for all efficacy endpoints. 158 and 147 patients in the nesiritide and placebo groups, respectively, were not MITT population eligible or didn't have outcome measure of interest.
Measure: Number; unit: Participants
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3406 | 3430
Participants
  Markedly Better | 449 | 418
  Moderately Better | 962 | 965
  Minimally Better | 1154 | 1186
  No Change | 751 | 785
  Minimally Worse | 42 | 49
  Moderately Worse | 17 | 11
  Markedly Worse | 31 | 16
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p = 0.318, Van Elteren test; Controlled for region

5. Secondary Outcome: Overall Well-Being Self-Assessment at 24 Hours After Initiation of Study Drug
Description: Overall well-being was measured by patient self-assessed Likert scale at 24 hours after study drug initiation. The Likert scale is a 7-point ordinal categorical scale (the 7 categories are markedly better, moderately better, minimally better, unchanged, minimally worse, moderately worse, and markedly worse.)
Time Frame: 24 hours after study drug initiation
Population: The modified intent-to-treat (MITT) population consisted of all randomized patients who received any amount of study medication and was the primary analysis population for all efficacy endpoints. 200 and 194 patients in the nesiritide and placebo groups, respectively, were not MITT population eligible or didn't have outcome measure of interest.
Measure: Number; unit: Participants
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3364 | 3383
Participants
  Markedly Better | 913 | 843
  Moderately Better | 1297 | 1311
  Minimally Better | 761 | 798
  No Change | 310 | 331
  Minimally Worse | 31 | 52
  Moderately Worse | 16 | 22
  Markedly Worse | 36 | 26
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p = 0.018, Van Elteren test; Controlled for region

6. Secondary Outcome: Composite of Persistent or Worsening Heart Failure and All-Cause Mortality
Description: Clinical manifestations of worsening or persistent decompensated heart failure were defined by at least one of the following: new, persistent or worsening: dyspnea, orthopnea, paroxysmal nocturnal dyspnea, edema, pulmonary basilar rales/crackles, jugular venous distension, renal hypoperfusion with no other apparent cause, or radiologic evidence of worsening heart failure. And was also defined by a new therapy specifically for the treatment of worsening or persistent decompensated heart failure.
Time Frame: Randomization to hospital discharge (up to Day 30)
Population: The modified intent-to-treat (MITT) population consisted of all randomized patients who received any amount of study medication and was the primary analysis population for all efficacy endpoints. 105 and 115 patients in the nesiritide and placebo groups, respectively, were not MITT population eligible or didn't have outcome measure of interest.
Measure: Number; unit: Participants
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3459 | 3462
Participants | 147 | 165
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p = 0.295, Cochran-Mantel-Haenszel; Controlled for region; Risk Difference (RD) = -0.5, 95% CI 2-sided [-1.5 to 0.5]

7. Secondary Outcome: Number of Days Alive and Outside the Hospital
Time Frame: Randomization to Day 30
Population: The modified intent-to-treat (MITT) population consisted of all randomized patients who received any amount of study medication and was the primary analysis population for all efficacy endpoints. 182 and 188 patients in the nesiritide and placebo groups, respectively, were not MITT population eligible or didn't have outcome measure of interest.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3382 | 3389
Days | 20.9 (6.88) | 20.7 (7.05)
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p = 0.160, ANOVA; Controlled for region; Mean Difference (Net) = 0.2, Standard Error of Mean 0.17 — This analysis excluded subjects who were lost to follow-up, or withdrawal of consent before Day 30, or whose Day 30 visit occurred prior to Day 30

8. Secondary Outcome: Composite of Cardiovascular Rehospitalization and Cardiovascular Mortality
Time Frame: Randomization to Day 30
Population: The modified intent-to-treat (MITT) population consisted of all randomized patients who received any amount of study medication and was the primary analysis population for all efficacy endpoints. 141 and 162 patients in the nesiritide and placebo groups, respectively, were not MITT population eligible or didn't have outcome measure of interest.
Measure: Number; unit: Participants
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3423 | 3415
Participants | 372 | 402
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p = 0.238, Cochran-Mantel-Haenszel; Controlled for region; Risk Difference (RD) = -0.9, 95% CI 2-sided [-2.4 to 0.6] — For subjects with a Day 30 visit prior to Day 30, information from their Day 180 visit, if available, was used to impute the mortality and rehospitalization status at Day 30

9. Other Pre Specified Outcome: All-Cause Mortality Through Day 30
Description: All deaths were adjudicated by an independent Clinical Events Committee.
Time Frame: Randomization to Day 30
Population: The safety population consisted of all randomized patients who received any amount of study medication. For all safety analyses, patients were analyzed according to the treatment actually received. 66 and 68 patients in the nesiritide and placebo groups, respectively, were not included in the safety population.
Measure: Number; unit: Participants
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3498 | 3509
Participants | 126 | 141

10. Other Pre Specified Outcome: All-Cause Mortality Through Day 180
Description: All deaths were adjudicated by an independent Clinical Events Committee.
Time Frame: Randomization to Day 180
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3498 | 3509
Participants | 429 | 447

11. Other Pre Specified Outcome: Cardiovascular Mortality Through Day 30
Description: All deaths were adjudicated by an independent Clinical Events Committee (CEC) and the cardiovascular deaths were classified by the CEC based on the primary causes.
Time Frame: Randomization to Day 30
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3498 | 3509
Participants
  Total Cardiovascular Deaths | 112 | 124
  Worsening Heart Failure | 68 | 80
  Myocardial Infarction | 4 | 0
  Sudden Cardiac Death | 20 | 23
  Other Cardiovascular Cause | 11 | 10
  Presumed Cardiovascular Cause | 9 | 11

12. Other Pre Specified Outcome: Number of Patients With Renal Impairment
Description: Renal impairment was defined as a greater than 25% decrease from baseline in the Modification of Diet in Renal Disease calculated glomerular filtration rate.
Time Frame: Study drug initiation to Day 30
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 3498 | 3509
Participants | 1032 | 968
Statistical Analysis 1: Comparison: Nesiritide vs Placebo; Test type: Superiority or Other; p = 0.109, Cochran-Mantel-Haenszel; Controlled for region; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.98 to 1.21]

ADVERSE EVENTS:
Arm/Group | Nesiritide | Placebo
Serious Adverse Events (participants affected / at risk) | 5/3498 | 2/3509
Other Adverse Events (participants affected / at risk) | 366/3498 | 364/3509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nesiritide (N=3498) | Placebo (N=3509)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Ischaemic Stroke (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nesiritide (N=3498) | Placebo (N=3509)
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Aortic Valve Stenosis (Cardiac disorders) | 1 | 0
Arrhythmia Supraventricular (Cardiac disorders) | 6 | 4
Atrial Fibrillation (Cardiac disorders) | 46 | 33
Atrial Flutter (Cardiac disorders) | 3 | 2
Atrial Septal Defect (Cardiac disorders) | 1 | 0
Atrial Tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 7 | 7
Cardiac Arrest (Cardiac disorders) | 16 | 10
Cardiac Tamponade (Cardiac disorders) | 1 | 0
Congestive Cardiomyopathy (Cardiac disorders) | 0 | 1
Electromechanical Dissociation (Cardiac disorders) | 1 | 0
Endocarditis (Cardiac disorders) | 2 | 1
Fluid Overload (Cardiac disorders) | 0 | 1
Hepatic Congestion (Cardiac disorders) | 1 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral Valve Incompetence (Cardiac disorders) | 0 | 1
Mitral Valve Prolapse (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 3
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Subacute Endocarditis (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 11 | 8
Ventricular Septal Defect (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 23 | 30
Carcinoid Tumour of the Appendix (Endocrine disorders) | 1 | 0
Diabetes Mellitus (Endocrine disorders) | 0 | 1
Diabetes Mellitus Inadequate Control (Endocrine disorders) | 1 | 1
Diabetic Neuropathy (Endocrine disorders) | 0 | 1
Hyperglycaemia (Endocrine disorders) | 2 | 2
Hypoglycaemia (Endocrine disorders) | 5 | 8
Hypothyroidism (Endocrine disorders) | 1 | 0
Blindness Transient (Eye disorders) | 1 | 0
Vision Blurred (Eye disorders) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 5 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2
Anal Abscess (Gastrointestinal disorders) | 1 | 0
Appendicitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Faeces Discoloured (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 3 | 2
Gastroenteritis Viral (Gastrointestinal disorders) | 0 | 2
Gastrointestinal Erosion (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 1
Rectal Abscess (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 1 | 2
Device Dislocation (General disorders) | 0 | 1
Device Related Infection (General disorders) | 1 | 0
Device Related Sepsis (General disorders) | 2 | 0
Hypothermia (General disorders) | 0 | 1
Infusion Site Extravasation (General disorders) | 2 | 0
Medical Device Complication (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Sudden Cardiac Death (General disorders) | 0 | 2
Sudden Death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 2 | 2
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic Encephalopathy (Hepatobiliary disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Hepatocellular Injury (Hepatobiliary disorders) | 1 | 0
Guillain-Barre Syndrome (Immune system disorders) | 0 | 1
Transfusion Reaction (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Enterococcal Bacteraemia (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 6 | 5
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 2
Staphylococcal Infection (Infections and infestations) | 3 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0
Streptococcal Sepsis (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 1
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Antimicrobial Susceptibility Test Resistant (Investigations) | 0 | 1
Blood Creatinine Increased (Investigations) | 2 | 0
Blood Glucose Increased (Investigations) | 0 | 1
Catheter Culture Positive (Investigations) | 0 | 1
Fibrin D Dimer Increased (Investigations) | 1 | 0
Gastric Ph Decreased (Investigations) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 1
International Normalised Ratio Increased (Investigations) | 0 | 2
Prostatic Specific Antigen Increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 6
Gout (Metabolism and nutrition disorders) | 2 | 2
Hyperbilirubinaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis Bacterial (Musculoskeletal and connective tissue disorders) | 1 | 0
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Sprain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lower Limb Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Patella Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft Tissue Infection (Musculoskeletal and connective tissue disorders) | 0 | 1
Colonic Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional State (Nervous system disorders) | 4 | 2
Convulsion (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Loss of Consciousness (Nervous system disorders) | 1 | 0
Unresponsive to Stimuli (Nervous system disorders) | 1 | 0
Acute Psychosis (Psychiatric disorders) | 1 | 0
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Failure to Thrive (Psychiatric disorders) | 0 | 2
Mental Status Changes (Psychiatric disorders) | 4 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Bladder Neoplasm (Renal and urinary disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal Artery Stenosis (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0
Ureteric Haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 1
Urinary Tract Infection (Renal and urinary disorders) | 1 | 7
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0
Urosepsis (Renal and urinary disorders) | 1 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breast Cancer (Reproductive system and breast disorders) | 1 | 0
Endometrial Cancer (Reproductive system and breast disorders) | 0 | 1
Orchitis (Reproductive system and breast disorders) | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Bronchitis Bacterial (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Eosinophilic Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxic Encephalopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infective Exacerbation of Chronic Obstructive Airways Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lobar Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lower Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Cancer Metastatic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Neoplasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Neoplasm Malignant (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Mediastinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinum Neoplasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Musculoskeletal Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Non-Cardiac Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 22 | 18
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Bacterial (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Mycoplasmal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Staphylococcal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acarodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2
Cellulitis (Skin and subcutaneous tissue disorders) | 4 | 2
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic Foot Infection (Skin and subcutaneous tissue disorders) | 0 | 1
Gangrene (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous Haematoma (Skin and subcutaneous tissue disorders) | 0 | 1
Abdominal Wall Haematoma (Vascular disorders) | 0 | 2
Acute Coronary Syndrome (Vascular disorders) | 1 | 0
Angina Pectoris (Vascular disorders) | 2 | 8
Angina Unstable (Vascular disorders) | 1 | 3
Aortic Aneurysm (Vascular disorders) | 0 | 1
Aortic Dissection (Vascular disorders) | 2 | 0
Aortic Stenosis (Vascular disorders) | 1 | 0
Arterial Haemorrhage (Vascular disorders) | 0 | 2
Bleeding Varicose Vein (Vascular disorders) | 0 | 1
Cardiogenic Shock (Vascular disorders) | 14 | 16
Catheter Site Haemorrhage (Vascular disorders) | 1 | 0
Cerebellar Haemorrhage (Vascular disorders) | 0 | 1
Cerebrovascular Accident (Vascular disorders) | 1 | 0
Colitis Ischaemic (Vascular disorders) | 1 | 0
Coronary Artery Disease (Vascular disorders) | 1 | 5
Deep Vein Thrombosis (Vascular disorders) | 4 | 3
Dizziness (Vascular disorders) | 0 | 4
Duodenal Ulcer Haemorrhage (Vascular disorders) | 1 | 0
Embolic Stroke (Vascular disorders) | 2 | 1
Embolism (Vascular disorders) | 0 | 1
Femoral Artery Occlusion (Vascular disorders) | 1 | 0
Gastrointestinal Haemorrhage (Vascular disorders) | 4 | 8
Haematemesis (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 1 | 1
Haemorrhagic Anaemia (Vascular disorders) | 0 | 1
Haemorrhagic Stroke (Vascular disorders) | 3 | 4
Haemorrhoidal Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 2
Hypoperfusion (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 6 | 10
Iliac Artery Embolism (Vascular disorders) | 1 | 0
Iliac Artery Thrombosis (Vascular disorders) | 0 | 1
Infusion Site Phlebitis (Vascular disorders) | 1 | 0
Intracardiac Thrombus (Vascular disorders) | 1 | 1
Ischaemic Cerebral Infarction (Vascular disorders) | 0 | 1
Ischaemic Hepatitis (Vascular disorders) | 0 | 1
Ischaemic Stroke (Vascular disorders) | 11 | 20
Lower Gastrointestinal Haemorrhage (Vascular disorders) | 1 | 0
Melaena (Vascular disorders) | 0 | 1
Myocardial Infarction (Vascular disorders) | 19 | 15
Myocardial Ischaemia (Vascular disorders) | 2 | 0
Orthostatic Hypotension (Vascular disorders) | 3 | 1
Peptic Ulcer Haemorrhage (Vascular disorders) | 0 | 1
Peripheral Embolism (Vascular disorders) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 1
Post Procedural Haematoma (Vascular disorders) | 0 | 2
Post Procedural Haemorrhage (Vascular disorders) | 0 | 1
Presyncope (Vascular disorders) | 0 | 5
Raynaud's Phenomenon (Vascular disorders) | 0 | 1
Rectal Haemorrhage (Vascular disorders) | 4 | 3
Retroperitoneal Haemorrhage (Vascular disorders) | 1 | 1
Septic Shock (Vascular disorders) | 3 | 3
Shock (Vascular disorders) | 0 | 1
Small Intestinal Haemorrhage (Vascular disorders) | 0 | 1
Subarachnoid Haemorrhage (Vascular disorders) | 1 | 0
Syncope (Vascular disorders) | 6 | 5
Systemic Inflammatory Response Syndrome (Vascular disorders) | 0 | 1
Thrombophlebitis Superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Transient Ischaemic Attack (Vascular disorders) | 2 | 4
Upper Gastrointestinal Haemorrhage (Vascular disorders) | 4 | 2

LIMITATIONS AND CAVEATS:
Only summary counts of deaths by group are provided for other pre-specified endpoints "All-cause mortality through Day 30" and "All-cause mortality through Day 180." Formal statistical comparisons were not planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Executive and Steering Committees is responsible for the creation, review, and submission of publications and presentations after study completion. The Investigator agrees that all data are the property of the Sponsors and subject to confidentiality and use restrictions until results are presented in the public domain. Publications or presentations must be submitted to the Sponsors and necessary committees for review before publication, public dissemination, or review by a third-parties.